CLINICAL TRIAL: NCT06361108
Title: A Phase I, Randomized, Double-Blind, Placebo Controlled MAD Study to Assess the Safety, Tolerability, PKs and Efficacy of Topical Application of YJ001 for Spray Use in Patients With DPNP
Brief Title: MAD Study to Assess the Safety, Tolerability, PKs and Efficacy of YJ001 for Spray Use in Patients With DPNP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Hanmai Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YJ001-103
Record Dates: First submitted 2024-03-19; First posted 2024-04-11 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Diabetes; Diabetic Peripheral Neuropathic(DPN); Diabetic Peripheral Neuropathic Pain(DPNP)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded with regard to the study treatment that subjects receive,without the investigator, the sponsor, or the subjects being aware of wether YJ001 or the placebo is administered. All decisions concerning dose escalation will be made in a blinded manner by the safety review committee.
  The Safety Review Committee (SRC), comprised of the Principal Investigator, Medical Monitor, and Sponsor's qualified designee, will convene after completion of each cohort to evaluate available safety, PK, and other relevant data.
  The SRC will determine whether to proceed to the next planned dose level, continue with the study and add additional safety evaluations, expand the number of subjects at the current level, reduce the dose, or stop the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort M1 (10active, 2 placebo) (Experimental): 296 mg/administration
  Interventions: Drug: YJ001 for Spray Use; Drug: Placebo of YJ001 for Spray Use
- Cohort M2 (10 active, 2 placebo) (Experimental): 414 mg/administration
  Interventions: Drug: YJ001 for Spray Use; Drug: Placebo of YJ001 for Spray Use

INTERVENTIONS:
Drug: YJ001 for Spray Use — Granules for spray use; Preparation of Dosing Solution: Reconstitute with sterile water (50ml)
Drug: Placebo of YJ001 for Spray Use — Inactive Ingredient: Sterile water; Preparation of Dosing Solution: 50ml Sterile water

SUMMARY:
This Phase I, randomized, double-blind and placebo controlled study is to evaluate the safety, tolerability, and PK, and to preliminarily assess the efficacy of topically administered YJ001 in a multiple-ascending dose (MAD) fashion in the patients with DPNP. The study will be conducted at a single study center.

In this study, 2 cohorts (N=24, 12 subjects for each cohort), each cohort will consist of 10 active and 2 placebo, with approximately equal numbers of male and female subjects.

Each subject will be administered a single dose of YJ001 as multiple sprays topically on both feet and below the ankle in the morning on Day 1 and Day 2, and will be administered as twice daily doses once in the morning and the other in the evening (with an interval of 11 to 13 h) from Day 3 through Day 11.

DETAILED DESCRIPTION:
This Phase I, randomized, double-blind and placebo controlled study is to evaluate the safety, tolerability, and PK, and to preliminarily assess the efficacy of topically administered YJ001 in a multiple-ascending dose (MAD) fashion in the patients with DPNP between ages of 18 to 80 years. The study will be conducted at a single study center.

In this study, 2 cohorts (N=24, 12 subjects for each cohort), the doses of which are 296 mg/administration (Cohort M1) and 414 mg/administration (Cohort M2), are planned. Each cohort will enroll approximately equal numbers of male and female subjects. The administration area is set as 450 cm2 (both feet). Each subject will be administered a single dose of YJ001 as multiple sprays (16 sprays/foot for Cohort M1, and 12 sprays/foot for Cohort M2) topically on both feet and below the ankle in the morning on Day 1 and Day 2, and will be administered as twice daily doses once in the morning and the other in the evening (with an interval of 11 to 13 h) from Day 3 through Day 11.

Each cohort will consist of 12 subjects (10 active; 2 placebo), with approximately equal numbers of male and female subjects.

Each cohort will be evaluated separately for safety and PK to allow for dose escalation based on stopping criteria per protocol. The Safety Review Committee (SRC), comprised of the Principal Investigator, Medical Monitor, and Sponsor's qualified designee, will convene after completion of each cohort to evaluate available safety, PK, and other relevant data. The decision whether to escalate the dose will be made for a completed cohort based on available safety data through Day 17 (5 days post the last dose), and blinded PK data [maximum observed plasma concentration (Cmax,ss) and area under the concentration-time curve through the first 48 hours post the last dose (AUC0-48h,ss)]. The SRC will determine whether to proceed to the next planned dose level, continue with the study and add additional safety evaluations, expand the number of subjects at the current level, reduce the dose, or stop the study.

Subjects will be screened between Day -28 through Day -7, rate the scores on Numeric Rating Scale (NRS) twice daily (once in the morning and the other in the evening) from Day -7 to Day -1, and will be admitted to the clinic on Day-1. Subjects will be housed within the clinic from Day -1 through Day 17 and will be discharged on Day 17 after all scheduled study procedures have been completed. If necessary, subjects will receive a telephone follow-up 2 days post discharge for documentation of any adverse event or concomitant medication.

Safety,Pharmacokinetics and Efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between the ages of 18 to 80 years at screening, both inclusive.
* Subjects voluntarily consenting for participation in the study and having signed informed consent document. Subjects are required to understand verbal and/or written English or any other language in which a certified translation of the informed consent is available.
* Body mass index (BMI) between 19 to 42 kg/m2 (both inclusive) at screening, calculated as weight (kg)/height2 (m2). Subjects must have two feet. Each foot must have five digits. Each foot must have at least total surface area of 450 cm2 measured from below the ankle to the toes including both dorsum and plantar areas.
* The subject is diagnosed with Type 1 or Type 2 diabetes, and has a history of DPNP for at least 3 months based on participant report or medical history.
* The subject should have a glycemic control that has been optimized and has been stable for at least 3 months prior to randomization. The subject has used a stable regimen of antidiabetic agents (oral) and/or insulin for at least 3 months before screening.
* Glycated hemoglobin (HbA1c) ≤ 10% at screening.
* Participants who have a weekly mean score of at least 4 based upon the daily mean scores using 11-point Numeric Rating Scale (NRS) in the daily diary (rated twice daily, once in the morning and the other in the evening) from Day -7 through Day 1 (should be calculated from records 7 days immediately prior to study drug administration).
* Males must not donate sperm until 90 days after last dose of study drug and must be willing to use a condom during heterosexual activity for up to 90 days after the application of the study drug.
* Females must be either postmenopausal for at least 1 year, surgically sterile (bilateral tubal ligation [including clip, cauterization methods and coil], bilateral oophorectomy or hysterectomy, and needs to be confirmed follicle-stimulating hormone [FSH] level >40 IU/L), or of childbearing potential either practicing true abstinence or practicing 2 effective means of contraception for at least 4 weeks prior to randomization, and until 28 days after study drug administration:

  1. Intrauterine device (IUD) or IUD hormone-releasing system.
  2. Combined estrogen and progestogen containing hormonal contraception (oral, intravaginal, or transdermal) associated with inhibition of ovulation.
  3. Progesterone-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation.
  4. Intrauterine hormone-releasing system.
  5. Double-barrier method (condoms, contraceptive sponge, diaphragm, or vaginal ring with spermicide).
* Able and willing to comply with all study requirements.

Exclusion Criteria:

* Current participation in another investigational drug or device study or treated with an investigational drug within 30 days or 5 half-lives, whichever is longer, before dosing.
* History of clinically significant drug, food allergy, skin allergy, or sensitivity to drugs of the same class (e.g., 5-aminosalicylic acid, sulfasalazine, and salicylates) or known hypersensitivity to YJ001 or any of its components.
* History of asthma. Adults with history of benign (resolved) childhood asthma may be included.
* Any subject who suffers severe peripheral vascular disease (e.g., intermittent claudication) at screening, and is not suitable to be involved in the study as per investigator evaluation.
* Any subject who suffers severe cardiovascular and cerebrovascular disease (e.g., severe arrhythmia, heart failure, myocardial infarction, unstable angina pectoris, atherosclerosis, stroke, sequela of stroke, etc.), severe gastrointestinal tract disease or other serious disease (e.g., cancer) which, in the opinion of the Investigator, would prevent the subject from fully participating in the study.
* Any subject who suffers chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) or multifocal motor neuropathy (MMN).
* Any subject who has a history of moderate to severe depression, obvious neurological or mental disorder not related to neuropathic pain but may interfere with rating of pain, as well as poly neuropathy, numbness, feeling of pins and needles and weakness in extremities, other serious pain cannot be clearly differentiated from or conditions that may interfere with rating of neuropathic pain. Subjects with weakness but w/o sensory complaints may be included.
* Any other medical, psychological, or social condition which, in the opinion of the Investigator, would prevent the subject from fully participating in the study, would represent a concern for study compliance, or would constitute a safety concern to the subject.
* Any subject who has suffered one or more severe hypoglycemia event (defined as neurofunctional hypoglycemia that needs third-party assistance) within 6 months prior to screening.
* Pain scores < 3 on the NRS over twice during the one-week run-in period.
* Any subject with unstable or poorly controlled abnormality in blood pressure or lipid (blood pressure ≥ 160 mmHg/95 mmHg, total cholesterol ≥ 6.2 mmol/L, and/or triglyceride ≥ 6.3 mmol/L) at screening.
* Any subject with abnormal renal function, estimated glomerular filtration rate (eGFR)<60 mL/min/1.73 m2.

eGFR=186×Scr^-1.154×Age^-0.203×(0.742 for Female)

* Any subject with abnormal liver function, liver enzymes (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) greater than 2 times upper limit of normal.
* Consumed 8 units or more of alcoholic beverages per week for women or 15 units or more of alcoholic beverages per week for men at any time in the 6 months before dosing (1 unit of ethanol is equivalent to 12 ounces of beer, 5 ounces of wine, or 1.5 ounces of spirits) or history of drug or alcohol abuse within the 6 months before dosing or evidence of such abuse as indicated by inquiry, medical history or the laboratory assays conducted during screening. Any subject who has past history of heavy drinking or alcoholism.
* Any subject who consumes more than 5 cigarettes per day within 30 days before study drug dosing or who cannot stop using any tobacco- or nicotine-containing product during the duration of the trial.
* Positive screening or check-in alcohol/drugs of abuse/cotinine screen.
* Positive test results for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Screening. SARS-CoV-2 testing will be either antigen, nasopharyngeal (NP) or nasal swab polymerase chain reaction (PCR) performed at Day -1, and in accordance with Centers for Disease Control and Prevention (CDC), FDA and local health authorities at the time of enrollment for this study. Participants not willing to comply with the investigational site's Coronavirus Disease 2019 (COVID 19) policy.
* Female volunteers who are pregnant or lactating.
* Have a significant acute illness within 7 days prior to study drug administration or have had a major illness or hospitalization within 1 month prior to study drug administration.
* Systemic or topical use of aspirin or salicylic acid containing products or sulfasalazine/salicylic acid derivatives within 14 days of study drug dosing.
* Use of other prescription and non-prescription medications (with the exception of permitted concomitant medications, oral contraceptives, combined estrogen and progestogen containing hormonal contraception and progestogen-only hormonal contraception), such as blood thinners, or sucralfate or herbal preparations within 14 days or 5 half-lives (whichever is longer) before study drug dosing, or use of an over-the-counter medication, vitamins, or supplements (including fish liver oils) within 14 days before study drug dosing.
* Positive screen on Hepatitis B, Hepatitis C, or Human immunodeficiency virus (HIV) at the time of screening evaluations.
* History of blood donation of more than 500 mL in the last 2 months prior to screening.
* History or evidence of poor venous access.
* History of bleeding disorders.
* Any subject with foot ulcers and/or pedal oedema. Presence of skin disorders, tattoos, skin breakdown, or other skin conditions on either foot that may interfere with the objectives of the study (as per investigator evaluation).
* Use of any kind of topical lotions, sunscreen, heating pads/cooling pads on feet for at least 24 hours before study drug is administered and until End-of-Study.
* An employee of the study center or Sponsor or family member of a study center employee
* Unwilling to stay in the clinical unit for the required duration as per the protocol or consume the standard meal to be provided as per the protocol.
* Any subject considering or scheduled to undergo any surgical procedure from screening to at least 7 days post dose.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety Assessments - AEs | through study completion, an average of 1year
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)
Safety Assessments -Number of Participants With Abnormal Laboratory Values | through study completion, an average of 1year
  Observed values and changes in baseline of clinical safety laboratory parameters
Safety Assessments - Skin Reaction | through study completion, an average of 1year
  Administration site assessment

SECONDARY OUTCOMES:
Pharmacokinetics-AUC | Day 1-Day 28
  Pharmacokinetics of YJ001 and metabolites YJ001-A, YJ001-B, and YJ001-C will be evaluated.
  Area under the concentration-time curve (AUC)
Pharmacokinetics- Cmax | Day 1-Day 28
  Maximum observed plasma concentration post dose (Cmax)
Pharmacokinetics - tmax | Day 1-Day 28
  Time of maximum observed plasma concentration (tmax)
Pharmacokinetics - tlag | Day 1
  Time to first quantifiable plasma concentration (tlag)
Pharmacokinetics - t1/2 | Day 1-Day 28
  t1/2: Apparent terminal elimination half-life post dose
Pharmacokinetics - CLr/f,ss | Day 1 - Day 28
  CLr/f,ss: Apparent systemic clearance at steady-state
Efficacy evaluation indicator | Day -7 - Day 12
  Numerical Rating Scale (NRS): at screening, Day -7 to Day 12, NRS score from 0 to 10(integer), the higher score means the more pain
Efficacy evaluation indicators | Day 1 - Day 13
  Average Daily Sleep Interference score (ADSIS): Day 1 to Day 13, ADSIS score from 0 to 10(integer), the higher score means the sleep is more severely affected by pain
Efficacy evaluation indicators | Day -1, Day 12
  Short-form McGill Pain Questionnaire (SF-MPQ) total scores: Day -1, Day 12.
Efficacy evaluation indicators | Day -1, Day 7, Day 11
  Vibration perception thresholds (VPT) test (monofilament sensory test)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Scott Denham, Principal Investigator — 5430 Fredericksburg Rd, Suite 200, San Antonio Texas 78229
Locations (1):
- Clinical Trials of Texas,LLC, Fredericksburg, Texas, United States